CLINICAL TRIAL: NCT00965185
Title: Statin Therapy to Improve Inflammation and Atherosclerosis in HIV Patients
Brief Title: Statin Therapy to Improve Atherosclerosis in HIV Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Steven K. Grinspoon, MD, Professor of Medicine, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008-P-000257; R01HL095123 (NIH); HL 095123
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Results first posted 2015-02-26 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Cardiovascular Disease; HIV; Atherosclerosis; Inflammation; Statins, HMG-CoA; HIV Infections
Keywords: Cardiovascular Disease; HIV; Atherosclerosis; Inflammation; Statins; treatment experienced
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Inflammation; HIV Infections | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin (Experimental): 20 mg PO QD for the first 3 months, followed by 40 mg PO QD for the final 9 months.
  Interventions: Drug: atorvastatin
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: atorvastatin — 20 mg PO QD for the first 3 months, followed by 40 mg PO QD for the final 9 months.
  Arms: Atorvastatin
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
In HIV patients, statin therapy will attenuate plaque inflammation, thus, making plaques less vulnerable, will deter plaque progression, and improve endothelial function. In addition to known cholesterol-lowering and C-reactive protein lowering effects, immunomodulatory effects of statins will lead to a shift from pro-inflammatory monocyte and T cell subsets to less atherogenic subpopulations.

ELIGIBILITY:
Inclusion criteria:

1. Men and women age 18-60 with previously diagnosed HIV disease
2. Subclinical coronary artery disease as defined by presence of one or more plaque on coronary CTA without history of cardiac events or cardiac symptoms and no evidence of critical coronary stenosis. Target to background ratio (TBR) as determined by PET of > 1.6.
3. Stable anti-retroviral (ARV) therapy as defined by no changes in ARV regimen for >6 months
4. LDL-cholesterol >70 mg/dL and <130 mg/dL

Exclusion criteria:

1. History of acute coronary syndrome
2. Contraindication to statin therapy
3. Current statin use
4. AST or ALT two times greater than the upper limit of normal or receiving treatment for active liver disease
5. Renal disease or creatinine >1.5 mg/dL (given the risk of contrast nephropathy during CT angiography of the heart)
6. Infectious illness within past 3 months
7. Contraindication to beta-blocker (including moderate to severe asthma or heart block) or nitroglycerin use as these drugs are given as part of the standard cardiac CT protocol. Previous allergic reaction to beta blocker or nitroglycerin.
8. Body weight greater than 300 lbs due to CT scanner table limitations
9. Patients with previous allergic reactions to iodine-containing contrast media
10. Active illicit drug use
11. Patients who report any significant radiation exposure over the course of the year prior to randomization. Significant exposure is defined as:

    1. More than 2 percutaneous coronary interventions (PCI) within 12 months of randomization
    2. More than 2 myocardial perfusion studies within the past 12 months
    3. More than 2 CT angiograms within the past 12 months
    4. Any subjects with history of radiation therapy.
12. Patients already scheduled or being considered for a procedure or treatment requiring significant radiation exposure (e.g., radiation therapy, PCI, or catheter ablation of arrhythmia) within 12 months of randomization
13. Pregnancy or breastfeeding
14. Coronary artery luminal narrowing >70% seen on coronary CTA

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven K. Grinspoon, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Subramanian S, Tawakol A, Burdo TH, Abbara S, Wei J, Vijayakumar J, Corsini E, Abdelbaky A, Zanni MV, Hoffmann U, Williams KC, Lo J, Grinspoon SK. Arterial inflammation in patients with HIV. JAMA. 2012 Jul 25;308(4):379-86. doi: 10.1001/jama.2012.6698. PMID 22820791
- [Result] Lo J, Lu MT, Ihenachor EJ, Wei J, Looby SE, Fitch KV, Oh J, Zimmerman CO, Hwang J, Abbara S, Plutzky J, Robbins G, Tawakol A, Hoffmann U, Grinspoon SK. Effects of statin therapy on coronary artery plaque volume and high-risk plaque morphology in HIV-infected patients with subclinical atherosclerosis: a randomised, double-blind, placebo-controlled trial. Lancet HIV. 2015 Feb;2(2):e52-63. doi: 10.1016/S2352-3018(14)00032-0. Epub 2015 Jan 9. PMID 26424461
- [Derived] deFilippi C, Christenson R, Joyce J, Park EA, Wu A, Fitch KV, Looby SE, Lu MT, Hoffmann U, Grinspoon SK, Lo J. Brief Report: Statin Effects on Myocardial Fibrosis Markers in People Living With HIV. J Acquir Immune Defic Syndr. 2018 May 1;78(1):105-110. doi: 10.1097/QAI.0000000000001644. PMID 29419569

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled men and women with HIV disease, no history of cardiovascular disease or cardiac symptoms, and evidence of subclinical atherosclerosis at Massachusetts General Hospital in Boston, MA USA. The study was done from November, 2009 to January, 2014.
Pre-assignment Details: Of the 81 patients screened for the study, 40 completed the screening and were randomized to the two study arms.
Groups:
- Atorvastatin: Participants received 20 mg atorvastatin given orally daily for the first 3 months, followed by 40 mg atorvastatin daily for the final 9 months.
- Placebo: Participants received 20 mg placebo given orally daily for the first three months followed by 40 mg placebo daily for the next 9 months.
Period: Overall Study
Arm/Group | Atorvastatin | Placebo
Started | 19 | 21
1 Month Visit | 18 | 21
3 Month Visit | 18 | 21
6 Month Visit | 18 | 21
9 Month Visit | 18 | 21
Completed | 17 | 20
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin | Placebo | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 21 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (3.8) | 50.0 (5.6) | 51.1 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 15 | 17 | 32
Race/Ethnicity, Customized [Number; unit: participants]
  White | 13 | 13 | 26
  Black | 3 | 3 | 6
  Asian | 0 | 1 | 1
  Hispanic | 1 | 1 | 2
  More than one race | 2 | 1 | 3
  Unknown | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 19 | 21 | 40

OUTCOME MEASURES:

1. Primary Outcome: Coronary and Aortic Plaque Inflammation
Description: 12 month change in mean FDG-PET TBR (18-fluorodeoxyglucose positron emission tomography target-to-background ratio)
Time Frame: Measured at baseline and 1 year
Population: All participants with baseline and 12 month PET and CT scans of acceptable image quality to permit assessment of change over time in identical regions in serial scans. As a result, only a limited number of participants could be included.
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 10 | 11
ratio
  Mean FDG-PET TBR of aorta | 0.04 [-0.08 to 0.16] | -0.05 [-0.28 to 0.17]
  Mean FDG-PET TBR of most diseased segment of aorta | -0.03 [-0.17 to 0.12] | -0.06 [-0.25 to 0.13]

2. Secondary Outcome: Plaque Progression
Description: 12 month percent change in plaque volume
Time Frame: Measured at baseline and 1 year
Population: All available data were used.
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 17 | 20
Percent change
  12 month change in total plaque volume | -4.7 [-25.4 to 15.9] | 18.2 [1.5 to 59.9]
  12 month change in non-calcified plaque volume | -19.4 [-39.2 to 9.3] | 20.4 [-7.1 to 94.4]

3. Secondary Outcome: Endothelial Function
Description: Assessment of endothelial function was to be measured by endothelial vasodilator function.
Time Frame: 1 year
Population: Please note that we were unable to collect data for this outcome measure, entitled "Endothelial Function" due to equipment malfunction.
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Immune Function
Description: 12 month change in CD4 T-lymphocytes
Time Frame: Measured at baseline and 1 year
Population: All available data were used; data were not available for one subject who completed the study.
Measure: Mean (95% Confidence Interval); unit: cells per microliter
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 17 | 19
cells per microliter | 17 [-68 to 101] | 4 [-72 to 80]

5. Secondary Outcome: Lipid Profile
Description: 12 month change in lipid profile
Time Frame: Measured at baseline and 1 year
Population: All available data were used.
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 17 | 20
mmol/L
  12 month change in total cholesterol | -1.23 [-1.53 to -0.93] | 0.12 [-0.12 to 0.37]
  12 month change in HDL cholesterol | 0.02 [-0.11 to 0.16] | -0.04 [-0.17 to 0.09]
  12 month change in direct LDL | -1.00 [-1.38 to 0.61] | 0.30 [0.04 to 0.55]
  12 month change in triglycerides | -0.10 [-0.46 to 0.44] | 0.08 [-0.46 to 0.38]

6. Secondary Outcome: C-reactive Protein (CRP)
Description: 12 month change in Log CRP concentration
Time Frame: Measured at baseline and 1 year
Population: All available data were used.
Measure: Mean (95% Confidence Interval); unit: log(mg/L)
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 17 | 20
log(mg/L) | -0.3 [-0.6 to 0.0] | 0.1 [-0.2 to 0.3]

7. Secondary Outcome: Adipocytokines
Description: 12 month change in IL-6
Time Frame: Measured at baseline and 1 year
Measure: Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 17 | 20
pg/ml | -1.25 [-2.90 to 0.40] | 0.41 [-0.44 to 1.26]

8. Secondary Outcome: Liver Function Tests (LFTs)
Description: Number of participants with LFT abnormalities (greater than or equal to 3 times the upper limit of normal).
  For reference, the normal ranges for AST and ALT are shown below. Please note that the normal range for ALT at Labcorp changed over the course of the study. AST and ALT elevations were determined based on the normal range at the time the lab test was performed.
  ALT: 0-40 IU/L, 0-44 IU/L, or 0-55 IU/L AST: 0-40 IU/L
Time Frame: Measured at baseline, 1, 3, 6, 9, and 12 months
Population: All available data were used.
Measure: Number; unit: participants
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 19 | 21
participants | 3 | 2

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Atorvastatin | Placebo
Serious Adverse Events (participants affected / at risk) | 2/19 | 1/21
Other Adverse Events (participants affected / at risk) | 13/19 | 14/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin (N=19) | Placebo (N=21)
Hepatocellular carcinoma (Hepatobiliary disorders) | 0 (0) | 1 (1)
Fallopian tube cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Gastrointestinal virus induced dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atorvastatin (N=19) | Placebo (N=21)
Loose stools (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Muscle aches or cramps (Musculoskeletal and connective tissue disorders) | 6 | 5
Liver function test abnormalities (Hepatobiliary disorders) | 3 | 2 — Greater than or equal to three times upper limit of normal
Elevated fasting blood glucose (Metabolism and nutrition disorders) | 0 | 2 — Greater than 126 mg/dL
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Abdominal Pain (General disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
FDG-PET scan data was interpretable in only a limited subset of participants as a result of technical problems with manual co-registration (outcome 1). We were unable to collect data for endothelial function due to equipment malfunction (outcome 3).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No